CLINICAL TRIAL: NCT03727308
Title: A Prospective, Comparative Study of Clinical Outcomes Following Clinic-based Versus Self-use of Medical Abortion Using Mifepristone With Misoprostol
Brief Title: Study of Clinic-based Versus Self-use of Medical Abortion Pills
Acronym: MOC
Status: Completed | Type: Observational
Sponsor: Ipas (Other)
Collaborators: University of Health Science, Phnom Penh, Cambodia (Unknown)
Responsible Party: Sponsor
Other Study IDs: 0916 NECHR
Record Dates: First submitted 2018-10-28; First posted 2018-11-01 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-09

CONDITIONS: Induced Abortion; First Trimester Abortion; Misoprostol; Mifepristone
Keywords: medical abortion; self-use

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Women recruited from pharmacies: Investigators will enroll women seeking medical abortion pills without prescription from pharmacies.
  - Medical abortion pills sourced from pharmacies
  Interventions: Behavioral: Medical abortion pills sourced from pharmacies
- Women recruited from health clinics: Investigators will enroll women seeking medical abortion pills from clinics.
  - Medical abortion pills sourced from health clinics
  Interventions: Behavioral: Medical abortion pills sourced from health clinics

INTERVENTIONS:
Behavioral: Medical abortion pills sourced from pharmacies — One cohort using medical abortion pills sourced from pharmacies
  Groups: Women recruited from pharmacies
Behavioral: Medical abortion pills sourced from health clinics — One cohort using medical abortion pills sourced from health clinics
  Groups: Women recruited from health clinics

SUMMARY:
The goal of the study is to determine whether important clinical outcomes differ among women who access a combined medical abortion regimen from a pharmacy when compared with those who access it from a facility.

DETAILED DESCRIPTION:
Medical abortion with mifepristone and misoprostol within the first 10 weeks of pregnancy is safe and highly effective. Investigators aim to assess whether self-use of early (<9 weeks) medical abortion using mifepristone with misoprostol results in non-inferior rates of clinical outcomes when compared with clinic-based provision of medical abortion.

The investigators will prospectively recruit women who obtain medical abortion medication from pharmacies and clinics. Follow-up will occur by telephone during two phone calls within 30 days following the woman's abortion. A small number of adolescents will be recruited into a qualitative substudy.

ELIGIBILITY:
Inclusion Criteria:

Women are eligible for participation if they have purchased abortion medications (mifepristone-misoprostol) independently at a pharmacy or received them from a clinic for an unwanted pregnancy at less than 9 weeks since her last menstrual period (LMP). She must meet the following criteria:

* Be at least 15 years of age (may vary by country)
* Have a known LMP of less than 9 weeks
* No contraindications to medical abortion (list)
* Willing and able to give informed consent
* Have a mobile phone of which they are the independent user or be willing to be followed-up in person
* Willing to be contacted with questions about her abortion by telephone (optional in-person visit) at 3, 10-14 and 30 days following initial contact.
* Resident of country of study.

Exclusion criteria:

* Contraindications to mifepristone-misoprostol
* Age <15

Min Age: 15 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Women who are pregnant and seeking abortion in study sites.
Sampling Method: Non-Probability Sample
Enrollment: 4196 (Actual)
Dates: Start 2018-05-30 (Actual); Primary Completion 2021-06-02 (Actual); Study Completion 2021-06-02 (Actual)

PRIMARY OUTCOMES:
Need for additional treatment to complete abortion | Final assessment at 30 days following mifepristone administration
  The primary outcome of the study will be the need for additional treatment to complete the abortion (either aspiration or repeated misoprostol) following a woman taking the medical abortion pills.

SECONDARY OUTCOMES:
Serious complications/ morbidity | Final assessment at 30 days following mifepristone administration
  Number of participants who will have a complication such as hemorrhage requiring a blood transfusion, hospitalization, serious infection and undiagnosed (at the time of mifepristone) ectopic pregnancy.

OTHER OUTCOMES:
Uptake of postabortion contraception | 30 days
  Women's reported use of contraception (yes or no and method type) following medical abortion

CONTACTS AND LOCATIONS:
Overall Officials: Nathalie Kapp, MD, MPH, Principal Investigator — Ipas
Locations (2):
- University of Health Sciences, Phnom Penh, Cambodia
- Regional Institute for Population Studies, Accra, Ghana

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kapp N, Bawah AA, Agula C, Menzel JL, Antobam SK, Asuming PO, Eckersberger E, Pearson EE. Medical abortion in Ghana: A non-randomized, non-inferiority study of access through pharmacies compared with clinics. Contraception. 2024 Dec;140:110538. doi: 10.1016/j.contraception.2024.110538. Epub 2024 Jul 11. PMID 39002625